CLINICAL TRIAL: NCT00831922
Title: A Multicenter, Open Label, Randomized, Parallel-group Study to Evaluate the Efficacy of Oral AB1010 in Adult Patients With Active Rheumatoid Arthritis With Inadequate Response to at Least One Disease Modifying Anti Rheumatic Drugs (DMARD)
Brief Title: Efficacy of Oral AB1010 in Adult Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB04012
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; DMARD failure; ACR
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — masitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): masitinib (AB1010) 3 mg/kg/day
  Interventions: Drug: masitinib (AB1010)
- 2 (Experimental): masitinib (AB1010) 6 mg/kg/day
  Interventions: Drug: masitinib (AB1010)

INTERVENTIONS:
Drug: masitinib (AB1010) — 3 mg/kg/day
  Arms: 1
Drug: masitinib (AB1010) — 6 mg/kg/day
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the activity of 2 oral doses of AB1010 in subjects suffering from active RA who have shown an inadequate response to one DMARD including MTX or anti-TNF, after 3 months (12 weeks) of treatment.

The safety and efficacy will be evaluated on:

Rate of patients achieving ACR 20, 50, 70 and 90 DAS (disease activity score) after 3 months treatment ACRn after 3 months treatment Therapeutic maintenance of AB1010 at 3 months Quality of Life assessed by SF12 Health Assessment Questionnaire (HAQ) Clinical and biological safety Pharmacokinetic profile of AB1010

ELIGIBILITY:
Inclusion Criteria:

1. Meet American College of Rheumatology (ACR) criteria for RA
2. Have active RA
3. ACR functional class I-III
4. Disease onset at > 16 years of age
5. Disease duration of at least 6 months
6. Failure to one DMARD including methotrexate and anti-TNF alpha

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Inadequate bone marrow function
3. Current use of a DMARD within 4 weeks (or 5 half-lives, whichever is longer) of screening except for leflunomide which requires a specific wash-out
4. Any previous use of recombinant IL1-Ra
5. Current use of more than 1 non steroidal anti-inflammatory drug (NSAID) or change of dose of the NSAID within 4 weeks of baseline or NSAID use greater than the maximum recommended dose
6. Within 4 weeks before baseline, use of more than 10 mg/day of prednisone or equivalent or change in the dose of prednisone or equivalent, or having intra-articular corticosteroid injection or bolus intramuscular or intravenous treatment with corticosteroids (>20 mg prednisone or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-09; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
rate of patients achieving ACR 20, 50, 70 and 90 at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
DAS (disease activity score) at 12 weeks | 12 weeks
ACRn at 12 weeks | 12 weeks
improvement of quality of life assessed by SF12 at 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, MD, PhD, Principal Investigator — Hôpital Kremlin Bicêtre, France

REFERENCES:
- [Result] Tebib J, Mariette X, Bourgeois P, Flipo RM, Gaudin P, Le Loet X, Gineste P, Guy L, Mansfield CD, Moussy A, Dubreuil P, Hermine O, Sibilia J. Masitinib in the treatment of active rheumatoid arthritis: results of a multicentre, open-label, dose-ranging, phase 2a study. Arthritis Res Ther. 2009;11(3):R95. doi: 10.1186/ar2740. Epub 2009 Jun 23. PMID 19549290